CLINICAL TRIAL: NCT04527640
Title: Effects of Synbiotics Supplementation on the Concentration of the Uremic Toxin Indoxyl Sulfate, Symptoms of Constipation, and Constipation-related Quality of Life in End-stage Renal Disease Patients Undergoing Hemodialysis
Brief Title: Effects of Synbiotics Supplementation on the Uremic Toxin Indoxyl Sulfate Level and Constipation in End-stage Renal Disease Patients Undergoing Hemodialysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr. Aida Lydia, PhD, SpPD-KGH, Teaching Staff, Faculty of Medicine, Indonesia University; Head of Kidney & Hypertension Division, Faculty of Medicine, Indonesia University, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 20-07-0796
Record Dates: First submitted 2020-08-20; First posted 2020-08-26 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Constipation; End Stage Renal Disease on Dialysis
Keywords: Synbiotics; Indoxyl Sulfate; Constipation; Quality of life; Dysbiosis; End-Stage Renal Disease; Hemodialysis
MeSH Terms: conditions — Constipation; Dysbiosis; Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: This study is a double-blind, placebo-controlled, randomized clinical trial conducted on end-stage renal disease patients undergoing hemodialysis. Patients will be randomized into two arms: symbiotic and placebo. The study will take place in the hemodialysis unit of Dr. Cipto Mangunkusumo General Hospital in September 2020 to February 2021. A total of 60 participants will be recruited for the study (30 in each arm). Both investigators and patients will be blinded to the treatment, and blinding will be conducted by the pharmacy unit of Dr. Cipto Mangunkusumo General Hospital.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Masking is done for participants, care provider, and investigator. Masking is assigned by the pharmacy unit of Dr. Cipto Mangunkusumo Hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synbiotic Arm (Experimental): Patients receiving synbiotics: Lactobacillus acidophilus & Bifidobacterium longum 5x10^9 Colony Forming Unit (CFU) and Fructooligosaccharides (FOS) 60 mg, 2 capsules/day for 60 days
  Interventions: Dietary Supplement: Synbiotics containing Lactobacillus acidophilus & Bifidobacterium longum 5x10^9 CFU and FOS 60 mg
- Placebo Arm (Placebo Comparator): Patients receiving placebo capsules containing saccharum lactis (2 capsules/day for 60 days)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Synbiotics containing Lactobacillus acidophilus & Bifidobacterium longum 5x10^9 CFU and FOS 60 mg — Patients will undergo baseline examination including medical history and physical examination, blood samples will be collected for hemoglobin, WBC, platelet, urea, creatinine, albumin and indoxyl sulfate level. Patients will be asked to complete 2 questionnaires the PAC-SYM and PAC-QOL questionnaires, and will undergo food recall evaluations by a nutritionist. They will then be given 2 capsules of synbiotics per day for 30 days. After 1 month of intervention, the patients will be evaluated for food recall and side effects. Afterwards, the patients will receive 2 capsules of the same synbiotics per day for the next 30 days. After 2 months of intervention, the patients' history will be taken, they will be asked to complete the PAC-SYM and PAC-QOL questionnaires, undergo food recall examination, and side effects evaluation. Blood samples will be taken for indoxyl sulfate examination.
  Arms: Synbiotic Arm
Other: Placebo — Patients will undergo baseline examination including medical history and physical examination, blood samples will be collected for hemoglobin, WBC, platelet, urea, creatinine, albumin and indoxyl sulfate level. Patients will be asked to complete 2 questionnaires the PAC-SYM and PAC-QOL questionnaires, and will undergo food recall evaluations by a nutritionist. They will then be given 2 capsules of placebo per day for 30 days. After 1 month of intervention, the patients will be evaluated for food recall and side effects. Afterwards, the patients will receive 2 capsules of the same placebo per day for the next 30 days. After 2 months of intervention, the patients' history will be taken, they will be asked to complete the PAC-SYM and PAC-QOL questionnaires, undergo food recall examination, and side effects evaluation. Blood samples will be taken for indoxyl sulfate examination.
  Arms: Placebo Arm

SUMMARY:
This is a double-blind, placebo-controlled, randomized clinical trial conducted to evaluate the effects of synbiotics supplementation on the level of the uremic toxin indoxyl sulfate, symptoms of constipation, and constipation-related quality of life in end-stage renal disease patients undergoing hemodialysis.

DETAILED DESCRIPTION:
One of the most common gastrointestinal symptoms in end-stage renal disease patients undergoing hemodialysis is constipation, which is one of the risk factors of microbiota dysbiosis. One effect of dysbiosis is the increased level of a uremic toxin known as indoxyl sulfate. The accumulated concentration of indoxyl sulfate in end-stage renal disease patients undergoing hemodialysis is associated with inflammation and oxidative stress, which in turn increases the risk of cardiovascular event. Constipation and an increased risk of cardiovascular event is associated with low quality of life in chronic kidney disease patients undergoing hemodialysis.

Synbiotics administrations had become one of the many ways to improve gut dysbiosis as it is expected to lower the level of indoxyl sulfate and improve the symptoms of constipation and constipation-related quality of life. Although studies had investigated the role of probiotics/prebiotics/synbiotics, the role of synbiotics in lowering the concentration of the uremic toxin indoxyl sulfate remains inconclusive. Therefore, this study is conducted to demonstrate the benefits of synbiotics administration in lowering the concentration of indoxyl sulfate in end-stage renal disease patients undergoing hemodialysis, This is the first study in Indonesia investigating the effects of synbiotics supplementation in end-stage renal disease patients undergoing hemodialysis.

This study is a double-blind, placebo-controlled, randomized clinical trial conducted on end-stage renal disease patients undergoing hemodialysis. Patients will be divided into two arms: synbiotics and placebo. The study will take place in the hemodialysis unit of Dr. Cipto Mangunkusumo General Hospital in September 2020 to February 2021. A total of 60 participants will be recruited for the study (30 in each arm), who will be randomized into the synbiotic arm or the placebo arm. Both investigators and patients will be blinded to the treatment, and blinding will be conducted by the pharmacy unit of Dr. Cipto Mangunkusumo General Hospital.

Patients who had consented to participate will be assessed for medical history and physical examination. Food recall evaluation will also be performed by a nutritionist. Blood samples will be collected from the patient for laboratory examinations, including haemoglobin, white blood cells (WBC), platelet, urea, creatinine, albumin, and indoxyl sulfate. Patients will also be asked to complete two questionnaires: the Patient Assessment of Constipation Symptoms (PAC-SYM) questionnaire to assess the symptoms of constipation and the Patient Assessment of Constipation Quality of Life (PAC-QOL) questionnaire to assess constipation-related quality of life. After this, patients will be randomized into one of the two study arms. The data will serve as baseline data.

Patients will receive 2 capsules containing either synbiotics or placebo per day for the next 30 days. Afterwards, the patients will undergo examination to evaluate food recall and side effects. After evaluation, the patients will once again receive 2 capsules containing either synbiotics or placebo per day for the next 30 days, and after a total 2 months of interventions, will undergo examinations similar to that done in baseline examination.

The primary outcome of this study is the concentration of indoxyl sulfate in end-stage renal disease patients undergoing hemodialysis. Secondary outcomes include the symptoms of constipation and constipation-related quality of life in end-stage renal disease patients undergoing hemodialysis.

This study will be done according to the principles detailed in Helsinki declaration, Guideline for Good Clinical Practice from ICH Tripartite Guideline (ICH-GCP), and had been approved by the Ethical Committee of the Faculty of Medicine of Indonesia University.

ELIGIBILITY:
Inclusion Criteria:

* Aged more than 18 years old
* Had undergone hemodialysis twice a week for a minimum of 3 months, with each visit lasting 5 hours
* Had only undergone hemodialysis therapy (not peritoneal dialysis/kidney transplantation)
* No history of malignancy or undergoing chemotherapy/radiation therapy
* No history of autoimmune disease or consuming immunosuppressants
* No history of bowel resection
* Had never been diagnosed with Crohn's disease or ulcerative colitis

Exclusion Criteria:

* Patients whose hemodialysis schedule was changed from twice a week to three times a week
* Patients consuming prebiotics/probiotics/synbiotics within the past 3 weeks
* Patients experiencing infection or is consuming antibiotics
* Patients who are not willing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09-15 (Estimated); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Indoxyl Sulfate concentration | Through study completion, an average of 60 days
  Concentration of indoxyl sulfates in the subjects' blood samples

SECONDARY OUTCOMES:
Symptoms of constipation | Through study completion, an average of 60 days
  Constipation-related symptoms as assessed using Patient Assessment of Constipation Symptoms (PAC-SYM) questionnaire. Score will be assessed at the start and at the end of the study. Symptoms will be considered improved if there is a reduction of total score by 1 or more point(s).
Constipation-related quality of life | Through study completion, an average of 60 days
  Constipation-related quality of life as assessed using Patient Assessment of Constipation Quality of Life (PAC-QOL) questionnaire. Score will be assessed at the start and at the end of the study. Quality of life will be considered improved if there is a reduction of total score by 1 or more point(s).

CONTACTS AND LOCATIONS:
Overall Officials: Aida Lydia, MD, PhD, Principal Investigator — Indonesia University

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data

REFERENCES:
- [Background] Said S, Hernandez GT. The link between chronic kidney disease and cardiovascular disease. J Nephropathol. 2014 Jul;3(3):99-104. doi: 10.12860/jnp.2014.19. Epub 2014 Jul 1. PMID 25093157
- [Background] Hill NR, Fatoba ST, Oke JL, Hirst JA, O'Callaghan CA, Lasserson DS, Hobbs FD. Global Prevalence of Chronic Kidney Disease - A Systematic Review and Meta-Analysis. PLoS One. 2016 Jul 6;11(7):e0158765. doi: 10.1371/journal.pone.0158765. eCollection 2016. PMID 27383068
- [Background] Hasan M, Sutradhar I, Gupta RD, Sarker M. Prevalence of chronic kidney disease in South Asia: a systematic review. BMC Nephrol. 2018 Oct 23;19(1):291. doi: 10.1186/s12882-018-1072-5. PMID 30352554
- [Background] Khan YH, Mallhi TH, Sarriff A, Khan AH, Tanveer N. Prevalence of Chronic Kidney Disease in Asia: A Systematic Review of Population-Based Studies. J Coll Physicians Surg Pak. 2018 Dec;28(12):960-966. doi: 10.29271/jcpsp.2018.12.960. PMID 30501836
- [Background] Liyanage T, Ninomiya T, Jha V, Neal B, Patrice HM, Okpechi I, Zhao MH, Lv J, Garg AX, Knight J, Rodgers A, Gallagher M, Kotwal S, Cass A, Perkovic V. Worldwide access to treatment for end-stage kidney disease: a systematic review. Lancet. 2015 May 16;385(9981):1975-82. doi: 10.1016/S0140-6736(14)61601-9. Epub 2015 Mar 13. PMID 25777665
- [Background] Liu M, Li XC, Lu L, Cao Y, Sun RR, Chen S, Zhang PY. Cardiovascular disease and its relationship with chronic kidney disease. Eur Rev Med Pharmacol Sci. 2014 Oct;18(19):2918-26. PMID 25339487
- [Background] Tong J, Liu M, Li H, Luo Z, Zhong X, Huang J, Liu R, He F, Fu J. Mortality and Associated Risk Factors in Dialysis Patients with Cardiovascular Disease. Kidney Blood Press Res. 2016;41(4):479-87. doi: 10.1159/000443449. Epub 2016 Jul 20. PMID 27434642
- [Background] Kendrick J, Chonchol MB. Nontraditional risk factors for cardiovascular disease in patients with chronic kidney disease. Nat Clin Pract Nephrol. 2008 Dec;4(12):672-81. doi: 10.1038/ncpneph0954. Epub 2008 Sep 30. PMID 18825155
- [Background] Allon M. Evidence-based cardiology in hemodialysis patients. J Am Soc Nephrol. 2013 Dec;24(12):1934-43. doi: 10.1681/ASN.2013060632. Epub 2013 Oct 17. PMID 24136920
- [Background] Wong J, Piceno YM, DeSantis TZ, Pahl M, Andersen GL, Vaziri ND. Expansion of urease- and uricase-containing, indole- and p-cresol-forming and contraction of short-chain fatty acid-producing intestinal microbiota in ESRD. Am J Nephrol. 2014;39(3):230-237. doi: 10.1159/000360010. Epub 2014 Mar 8. PMID 24643131
- [Background] Zuvela J, Trimingham C, Le Leu R, Faull R, Clayton P, Jesudason S, Meade A. Gastrointestinal symptoms in patients receiving dialysis: A systematic review. Nephrology (Carlton). 2018 Aug;23(8):718-727. doi: 10.1111/nep.13243. PMID 29468835
- [Background] Sumida K, Yamagata K, Kovesdy CP. Constipation in CKD. Kidney Int Rep. 2019 Nov 13;5(2):121-134. doi: 10.1016/j.ekir.2019.11.002. eCollection 2020 Feb. PMID 32043026
- [Background] Zhang J, Huang C, Li Y, Chen J, Shen F, Yao Q, Qian J, Bao B, Yao X. Health-related quality of life in dialysis patients with constipation: a cross-sectional study. Patient Prefer Adherence. 2013 Jun 18;7:589-94. doi: 10.2147/PPA.S45471. Print 2013. PMID 23814466
- [Background] Ramezani A, Massy ZA, Meijers B, Evenepoel P, Vanholder R, Raj DS. Role of the Gut Microbiome in Uremia: A Potential Therapeutic Target. Am J Kidney Dis. 2016 Mar;67(3):483-98. doi: 10.1053/j.ajkd.2015.09.027. Epub 2015 Nov 15. PMID 26590448
- [Background] Claro LM, Moreno-Amaral AN, Gadotti AC, Dolenga CJ, Nakao LS, Azevedo MLV, de Noronha L, Olandoski M, de Moraes TP, Stinghen AEM, Pecoits-Filho R. The Impact of Uremic Toxicity Induced Inflammatory Response on the Cardiovascular Burden in Chronic Kidney Disease. Toxins (Basel). 2018 Sep 23;10(10):384. doi: 10.3390/toxins10100384. PMID 30249039
- [Background] Poesen R, Evenepoel P, de Loor H, Delcour JA, Courtin CM, Kuypers D, Augustijns P, Verbeke K, Meijers B. The Influence of Prebiotic Arabinoxylan Oligosaccharides on Microbiota Derived Uremic Retention Solutes in Patients with Chronic Kidney Disease: A Randomized Controlled Trial. PLoS One. 2016 Apr 21;11(4):e0153893. doi: 10.1371/journal.pone.0153893. eCollection 2016. PMID 27100399
- [Background] Rossi M, Klein K, Johnson DW, Campbell KL. Pre-, pro-, and synbiotics: do they have a role in reducing uremic toxins? A systematic review and meta-analysis. Int J Nephrol. 2012;2012:673631. doi: 10.1155/2012/673631. Epub 2012 Dec 19. PMID 23316359
- [Background] Nakabayashi I, Nakamura M, Kawakami K, Ohta T, Kato I, Uchida K, Yoshida M. Effects of synbiotic treatment on serum level of p-cresol in haemodialysis patients: a preliminary study. Nephrol Dial Transplant. 2011 Mar;26(3):1094-8. doi: 10.1093/ndt/gfq624. Epub 2010 Oct 7. PMID 20929916
- [Background] Natarajan R, Pechenyak B, Vyas U, Ranganathan P, Weinberg A, Liang P, Mallappallil MC, Norin AJ, Friedman EA, Saggi SJ. Randomized controlled trial of strain-specific probiotic formulation (Renadyl) in dialysis patients. Biomed Res Int. 2014;2014:568571. doi: 10.1155/2014/568571. Epub 2014 Jul 24. PMID 25147806
- [Background] Hyun HS, Paik KH, Cho HY. p-Cresyl sulfate and indoxyl sulfate in pediatric patients on chronic dialysis. Korean J Pediatr. 2013 Apr;56(4):159-64. doi: 10.3345/kjp.2013.56.4.159. Epub 2013 Apr 22. PMID 23646054
- [Background] Meijers BK, De Preter V, Verbeke K, Vanrenterghem Y, Evenepoel P. p-Cresyl sulfate serum concentrations in haemodialysis patients are reduced by the prebiotic oligofructose-enriched inulin. Nephrol Dial Transplant. 2010 Jan;25(1):219-24. doi: 10.1093/ndt/gfp414. Epub 2009 Aug 19. PMID 19692415
- [Background] Ramos CI, Armani RG, Canziani MEF, Dalboni MA, Dolenga CJR, Nakao LS, Campbell KL, Cuppari L. Effect of prebiotic (fructooligosaccharide) on uremic toxins of chronic kidney disease patients: a randomized controlled trial. Nephrol Dial Transplant. 2019 Nov 1;34(11):1876-1884. doi: 10.1093/ndt/gfy171. PMID 29939302
- [Background] Hida M, Aiba Y, Sawamura S, Suzuki N, Satoh T, Koga Y. Inhibition of the accumulation of uremic toxins in the blood and their precursors in the feces after oral administration of Lebenin, a lactic acid bacteria preparation, to uremic patients undergoing hemodialysis. Nephron. 1996;74(2):349-55. doi: 10.1159/000189334. PMID 8893154
- [Background] Takayama F, Taki K, Niwa T. Bifidobacterium in gastro-resistant seamless capsule reduces serum levels of indoxyl sulfate in patients on hemodialysis. Am J Kidney Dis. 2003 Mar;41(3 Suppl 1):S142-5. doi: 10.1053/ajkd.2003.50104. PMID 12612972
- [Background] Taki K, Takayama F, Niwa T. Beneficial effects of Bifidobacteria in a gastroresistant seamless capsule on hyperhomocysteinemia in hemodialysis patients. J Ren Nutr. 2005 Jan;15(1):77-80. doi: 10.1053/j.jrn.2004.09.028. PMID 15648012
- [Background] Sirich TL, Plummer NS, Gardner CD, Hostetter TH, Meyer TW. Effect of increasing dietary fiber on plasma levels of colon-derived solutes in hemodialysis patients. Clin J Am Soc Nephrol. 2014 Sep 5;9(9):1603-10. doi: 10.2215/CJN.00490114. Epub 2014 Aug 21. PMID 25147155
- [Background] Esgalhado M , Kemp JA , Azevedo R , Paiva BR , Stockler-Pinto MB , Dolenga CJ , Borges NA , Nakao LS , Mafra D . Could resistant starch supplementation improve inflammatory and oxidative stress biomarkers and uremic toxins levels in hemodialysis patients? A pilot randomized controlled trial. Food Funct. 2018 Dec 13;9(12):6508-6516. doi: 10.1039/c8fo01876f. PMID 30468238
- [Background] Rossi M, Johnson DW, Morrison M, Pascoe EM, Coombes JS, Forbes JM, Szeto CC, McWhinney BC, Ungerer JP, Campbell KL. Synbiotics Easing Renal Failure by Improving Gut Microbiology (SYNERGY): A Randomized Trial. Clin J Am Soc Nephrol. 2016 Feb 5;11(2):223-31. doi: 10.2215/CJN.05240515. Epub 2016 Jan 15. PMID 26772193
- [Background] Borges NA, Carmo FL, Stockler-Pinto MB, de Brito JS, Dolenga CJ, Ferreira DC, Nakao LS, Rosado A, Fouque D, Mafra D. Probiotic Supplementation in Chronic Kidney Disease: A Double-blind, Randomized, Placebo-controlled Trial. J Ren Nutr. 2018 Jan;28(1):28-36. doi: 10.1053/j.jrn.2017.06.010. Epub 2017 Sep 6. PMID 28888762
- [Derived] Lydia A, Indra TA, Rizka A, Abdullah M. The effects of synbiotics on indoxyl sulphate level, constipation, and quality of life associated with constipation in chronic haemodialysis patients: a randomized controlled trial. BMC Nephrol. 2022 Jul 22;23(1):259. doi: 10.1186/s12882-022-02890-9. PMID 35869437